CLINICAL TRIAL: NCT02632123
Title: Validation of the Risk Stratification Score in Idiopathic Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Western University, Canada (Other); University of Rome Tor Vergata (Other); University of Waterloo (Other)
Responsible Party: Sponsor
Other Study IDs: 10010803
Record Dates: First submitted 2015-12-13; First posted 2015-12-16 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: idiopathic pulmonary fibrosis; outcome; prognosis; survival; staging
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Development cohort: Patients newly diagnosed with idiopathic pulmonary fibrosis
- Validation cohort: Patients newly diagnosed with idiopathic pulmonary fibrosis

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is characterized by a poor prognosis, with a progressive decline in lung function and a considerable variability in the disease's natural history. Besides lung transplantation (LTx), the only available treatments are anti-fibrosing drugs, which have shown to slower the disease course. Therefore, predicting the prognosis is of pivotal importance to avoid treatment delays, which may be fatal for patients with a high risk of progression. Previous studies showed that a multi-dimensional approach is practical and effective to create a reliable prognostic score for IPF. In the RIsk Stratification scorE (RISE), physiological parameters, an objective measure of patient-reported dyspnea and exercise capacity are combined to capture different domains of the complex pathophysiology of IPF.

This is an observational, multi-centre, prospective cohort study. A development cohort and a validation cohort will be included. Patients newly diagnosed with IPF based on the ATS/ERS criteria and multi-disciplinary discussion will be included in the study. A panel of chest radiologists and lung pathologists will further assess eligibility. At the first visit (time of diagnosis), and every 4-months, MRCDS, pulmonary function tests (FEV1, FVC and DLCO), and 6MWD will be recorded and patients will be prospectively followed for 3 years. Comorbidities will be considered. The radiographic extent of fibrosis on HRCT will be recalculated at a 2-year interval. RISE, Gender-Age-Physiology, CPI and Mortality Risk Scoring System will be calculated at 4-month intervals. Longitudinal changes of each variable considered will be assessed. The primary endpoint is 3-year LTx-free survival from the time of diagnosis. Secondary endpoints include several, clinically-relevant information to ensure reproducibility of results across a wide range of disease severity and in concomitance of associated pulmonary hypertension, emphysema.

The present study aims at validating RISE as a simple, straightforward, inexpensive and reproducible tool to guide clinical decision making in IPF and potentially as an endpoint for future clinical trials.

DETAILED DESCRIPTION:
This is an observational, international, prospective cohort study including 2 large tertiary referral centres for interstitial lung disease (ILD)(London, Canada and Rome, Italy). Only patients newly diagnosed with IPF based on the American Thoracic Society/European Respiratory Society criteria and local multi-disciplinary discussion will be included in the study.

As a further inclusion step, for all patients who did not undergo a surgical lung biopsy (SLB), a panel of 3 chest radiologists with ILD expertise will examine each HRCT and patients will be included, if at least 2 out of 3 agree on a pattern of probable/definite UIP. For patients who underwent a SLB, a panel of 3 lung pathologists with ILD expertise will examine each biopsy and patients will be included, if at least 2 out of 3 agree on a pattern of probable/definite UIP.

All known causes of ILD (occupational, environmental, domestic exposures; drug-induced lung toxicity; connective tissue disease) will carefully excluded for the patient to be included in the study. Only patients newly diagnosed with IPF at participating centres will be included in the study. Comorbidities considered will include (associated pulmonary hypertension [APH], only if right heart catheterization[RHC]-proven), chronic obstructive pulmonary disease (COPD), coronary artery disease (CAD), left heart dysfunction (LHD), and sleep apnea (SA).

A development cohort and a validation cohort will be included in the study. In both cohorts. at the first visit (time of diagnosis) and at each subsequent visit at 4-month intervals, for a period of 3 years, Medical Research Council Dyspnea Score (MRCDS), pulmonary function tests (PFTs)(forced expiratory volume during the first second [FEV1], FVC and diffusing lung capacity for carbon monoxide [DLCO]), and 6MWD will be recorded. 6MWD % predicted will be calculated, as previously described.

The following events will be recorded in the study: death; lung transplant (LTx) referral; LTx; acute exacerbation (AEs); hospitalization for respiratory causes; start, stop and switch of anti-fibrotic therapy; start of supplemental home oxygen therapy; start and stop of physiotherapy program enrolments; progression of disease (see secondary endpoints).

The RISE will be first calculated, as previously described, on a scale from 1 to 3. However, a modified and improved version of the RISE will also be considered, both using the CALIPER-revised Composite Physiologic index (CPI) instead of the original version of CPI, and with a new 1 to 4 scale, which may allow for better stratification for mortality risk. If superior to the previous version of RISE, the modified version will be tested for validation.

Patients will be prospectively followed for a period of 3 years from the time of diagnosis and enrolment. PFTs and 6MWD will be obtained at 4 months intervals, at each visit at participating centres. All multi-dimensional scores will be calculated at 4-months intervals corresponding to each visit. A 2nd HRCT will be obtained at the 2-year visit, or sooner if clinically indicated, and as per clinicians' discretion. The HRCT fibrosis score will be then recalculated on the 2nd scan. Deaths, LTx, AEs and hospitalizations due to respiratory causes will be recorded. All protocol violations (missing visits, delayed visits, data not obtained at individual visits) will be systematically recorded. Every interruption or change in course of therapy, as well as initiation of supplemental home oxygen therapy will be recorded. When available, hemodynamic data from RHCs will be considered. Since 2D echocardiograms alone are unreliable in predicting the presence of APH in IPF, they will not be considered.

At the end of the study period, both baseline RISE and longitudinal changes of RISE will be tested as predictors of mortality. Other individual variables will also be tested as predictors of mortality, including age at the time of diagnosis, time between onset of symptoms and diagnosis (months), gender, body mass index, smoking history (pack-years), FVC, DLCO, 6MWD (meters and % predicted), HRCT visual fibrosis score at the time of diagnosis, and other multi-dimensional scores (Gender-Age-Physiology [GAP], CPI, Mortality Risk Scoring System [MRSS]). In the validation cohort, we will seek to confirm and validate results obtained in the development cohort.

PATIENT SELECTION Inclusion criteria A new diagnosis of IPF based on ATS/ERS criteria, confirmed by local multi-disciplinary discussion (MDD). A panel of 3 chest radiologists with ILD expertise will review each HRCT and patients will be included, if at least 2 out of 3 agree on a pattern of probable/definite UIP. A panel of 3 lung pathologists with ILD expertise will review each SLB and patients will be included, if at least 2 out of 3 agree on a pattern of probable/definite UIP.

Exclusion criteria ILD other than IPF Previous (rather than new) diagnosis of IPF Exclusion determined by the chest radiologists' or lung pathologists' panel Age <18 years Patient not able to provide informed consent

MRC dyspnea score, pulmonary function tests and 6-minute walk test Dyspnea, defined as "the unpleasant sensation of labored or difficult breathing" was rated by using the MRCDS, which specifically measures perceived respiratory disability24. This scale grades the effect of breathlessness on daily activities. PFTs and 6-minute walk test (6MWT) will be performed according to ERS/ATS guidelines and the ATS guidelines, respectively. A reference equation was used to calculate 6MWD percent predicted (% pred). The distance-saturation product will be considered.

High resolution chest CT scans A quantitative fibrosis score on HRCT will be obtained at the time of diagnosis and on the repeat HRCT. The score will be calculated as previously described12 by each of the chest radiologists, and the average of the scores will then be calculated. Interobserver variability will be evaluated. The presence and severity of coronary calcifications will be evaluated as absent, mild, moderate or severe.

Longitudinal follow-up After diagnosis, patients are seen at 4-month intervals, for a period of 3 years in both the development and validation cohort. At each visit, MRCDS, PFTs and 6MWT will be obtained. Patients may be seen more often at the clinician's discretion. After completion of the 3 years follow-up period, patients who are still alive without a LTx will continue to be followed regularly until required recruitment is completed, as long-term follow-up is part of secondary endpoints.

Statistical Analysis and sample size calculation Values will be expressed as mean ± standard deviation. The Kolmogorov-Smirnov test will be used for distribution analysis. Interobserver variability among chest radiologists and lung pathologists will be assessed with Weighted kappa coefficients29. Comparisons between survivors and non-survivors will be made with unpaired t-test or with the Mann-Whitney U-test, where appropriate. Variance inflation factors of the predicting variables included in RISE will be calculated to rule out the possibility of multicollinearity and demonstrate that the variables are truly independent30. The optimal cut-off value for different variables to endpoints will be assessed using receiver operating characteristics analysis. Cox proportional hazards regression analysis will used to identify significant variables predicting survival status. Results will be summarized as hazard ratios, representing the relative risk of dying as a result of a specific characteristic during the observation period. Variables selected via univariate analysis (p<0.05) will be evaluated in the multivariate Cox regression analysis. Once patients are listed for LTx, death and LTx become competing events. In order to account for the competing risks of LTx and death in a population of patients undergoing LTx assessment, the Fine-Gray competing risk regression analysis will also be used to identify significant variables predicting independent survival status. Results will be summarized as subdistribution hazard ratios, representing the relative risk of dying prior to LTx. Survival will be further evaluated using Kaplan-Meier curves and the log-rank test.

ELIGIBILITY:
Inclusion Criteria:

* A new diagnosis of IPF based on the American Thoracic Society/European Respiratory Society criteria (Am J Respir Crit Care Med 2018;198:e44-e68) and confirmed by a panel of expert chest radiologists and lung pathologists in the context of multi-disciplinary discussion.

Exclusion Criteria:

* Interstitial lung disease other than IPF
* Not a new diagnosis of IPF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly diagnosed with idiopathic pulmonary fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Survival | 3 years
  Primary outcome is lung-transplant-free 3-year survival since the time of diagnosis

SECONDARY OUTCOMES:
Subgroup analysis | 3 years
  Comparative analysis of RISE as predictor of LTx-free survival in subgroups stratified by age; gender; baseline lung function; baseline 6MWD; baseline extent of fibrosis on HRCT; time between onset of symptoms and diagnosis; presence of APH; presence of concomitant emphysema; presence of comorbidities (COPD, CAD, LHD, SA); participating site
Clinical progression | 3 years
  Clinical progression as a predictor of mortality, defined as either: absolute decline of FVC >10% pred; decline of 6-min walk distance >50 m; hospitalization for respiratory causes; LTx assessment; or death
Incidence of acute exacerbations | 3 years
  Incidence of acute exacerbations (AEs) of IPF and its predictors, if any.
Incidence of hospitalizations | 3 years
  Incidence of hospitalizations due to respiratory causes and its predictors, if any.
Results stratification by HRT pattern | 3 years
  LTx-free survival, incidence of AEs, incidence of hospitalizations, and time to progression of patients with HRCT pattern definite/probable for UIP vs. patients with indeterminate/inconsistent pattern. In this subanalysis, 2 groups of patients matched for age, gender, BMI, and extent of fibrosis at the time of diagnosis will be considered.
Results stratification by autoimmune markers | 3 years
  LTx-free survival, incidence of AEs, incidence of hospitalizations, and time to progression of patients with autoimmune markers (although not meeting criteria for interstitial pneumonia with autoimmune features vs. those without. In this subanalysis, 2 groups of patients matched for age, gender, BMI and extent of fibrosis at the time of diagnosis will be considered
Results stratification by concomitant emphysema | 3 years
  LTx-free survival, incidence of AEs, incidence of hospitalizations and time to progression of patients with concomitant emphysema vs. those without. In this subanalysis, 2 groups of patients matched for age, gender, BMI and extent of fibrosis at the time of diagnosis will be considered.
Results stratification by anti-fibrotic treatment | 3 years
  LTx-free survival, incidence of AEs, incidence of hospitalizations and time to progression of patients treated with pirfenidone vs. patients treated with nintedanib. In this subanalysis, 2 groups of patients matched for age, gender, BMI and extent of fibrosis at the time of diagnosis will be considered.
Results stratification by anti-fibrotic treatment switch | 3 years
  LTx-free survival, incidence of AEs, incidence of hospitalizations and time to progression of patients whose therapy was switched (from pirfenidone to nintedanib and viceversa). In this subanalysis, 2 groups of patients matched for age, gender, BMI and extent of fibrosis at the time of diagnosis will be considered.
6MWD m vs. % pred as predictors of mortality | 3 years
  6-min walk distance in meters vs. percent predicted as predictors of mortality.
Results on patient listed for lung transplant | 3 years
  Survival, incidence of AEs and time to progression on the LTx list of listed patients.
Time to progression in patients with initially non-clinically significant disease. | 3 year
  Time to clinical progression in patients who initially had non-clinically significant disease
Long-term follow-up | 5 years
  Long-term follow-up (beyond 3 years) of patients who are still alive without a LTx, until required recruitment is completed. This will include LTx-free survival, incidence of AEs, incidence of hospitalizations and time to progression.

CONTACTS AND LOCATIONS:
Locations (2):
- London Health Science Centre, London, Ontario, Canada
- Policlinico Tor Vergata, Rome, Lazio, Italy

REFERENCES:
- [Background] Martinez FJ, Collard HR, Pardo A, Raghu G, Richeldi L, Selman M, Swigris JJ, Taniguchi H, Wells AU. Idiopathic pulmonary fibrosis. Nat Rev Dis Primers. 2017 Oct 20;3:17074. doi: 10.1038/nrdp.2017.74. PMID 29052582
- [Background] Raghu G, Remy-Jardin M, Myers JL, Richeldi L, Ryerson CJ, Lederer DJ, Behr J, Cottin V, Danoff SK, Morell F, Flaherty KR, Wells A, Martinez FJ, Azuma A, Bice TJ, Bouros D, Brown KK, Collard HR, Duggal A, Galvin L, Inoue Y, Jenkins RG, Johkoh T, Kazerooni EA, Kitaichi M, Knight SL, Mansour G, Nicholson AG, Pipavath SNJ, Buendia-Roldan I, Selman M, Travis WD, Walsh S, Wilson KC; American Thoracic Society, European Respiratory Society, Japanese Respiratory Society, and Latin American Thoracic Society. Diagnosis of Idiopathic Pulmonary Fibrosis. An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline. Am J Respir Crit Care Med. 2018 Sep 1;198(5):e44-e68. doi: 10.1164/rccm.201807-1255ST. PMID 30168753
- [Background] Mura M, Porretta MA, Bargagli E, Sergiacomi G, Zompatori M, Sverzellati N, Taglieri A, Mezzasalma F, Rottoli P, Saltini C, Rogliani P. Predicting survival in newly diagnosed idiopathic pulmonary fibrosis: a 3-year prospective study. Eur Respir J. 2012 Jul;40(1):101-9. doi: 10.1183/09031936.00106011. Epub 2012 Jan 12. PMID 22241745
- [Background] Ley B, Collard HR, King TE Jr. Clinical course and prediction of survival in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2011 Feb 15;183(4):431-40. doi: 10.1164/rccm.201006-0894CI. Epub 2010 Oct 8. PMID 20935110
- [Background] Farrand E, Iribarren C, Vittinghoff E, Levine-Hall T, Ley B, Minowada G, Collard HR. Impact of Idiopathic Pulmonary Fibrosis on Longitudinal Health-care Utilization in a Community-Based Cohort of Patients. Chest. 2021 Jan;159(1):219-227. doi: 10.1016/j.chest.2020.07.035. Epub 2020 Jul 24. PMID 32717266
- [Background] Nathan SD, Albera C, Bradford WZ, Costabel U, du Bois RM, Fagan EA, Fishman RS, Glaspole I, Glassberg MK, Glasscock KF, King TE Jr, Lancaster L, Lederer DJ, Lin Z, Pereira CA, Swigris JJ, Valeyre D, Noble PW, Wells AU. Effect of continued treatment with pirfenidone following clinically meaningful declines in forced vital capacity: analysis of data from three phase 3 trials in patients with idiopathic pulmonary fibrosis. Thorax. 2016 May;71(5):429-35. doi: 10.1136/thoraxjnl-2015-207011. Epub 2016 Mar 11. PMID 26968970
- [Background] Collard HR, Ryerson CJ, Corte TJ, Jenkins G, Kondoh Y, Lederer DJ, Lee JS, Maher TM, Wells AU, Antoniou KM, Behr J, Brown KK, Cottin V, Flaherty KR, Fukuoka J, Hansell DM, Johkoh T, Kaminski N, Kim DS, Kolb M, Lynch DA, Myers JL, Raghu G, Richeldi L, Taniguchi H, Martinez FJ. Acute Exacerbation of Idiopathic Pulmonary Fibrosis. An International Working Group Report. Am J Respir Crit Care Med. 2016 Aug 1;194(3):265-75. doi: 10.1164/rccm.201604-0801CI. PMID 27299520
- [Background] Serajeddini H, Rogliani P, Mura M. Multi-dimensional Assessment of IPF Across a Wide Range of Disease Severity. Lung. 2018 Dec;196(6):707-713. doi: 10.1007/s00408-018-0152-4. Epub 2018 Aug 27. PMID 30151723
- [Background] Fisher JH, Al-Hejaili F, Kandel S, Hirji A, Shapera S, Mura M. Multi-dimensional scores to predict mortality in patients with idiopathic pulmonary fibrosis undergoing lung transplantation assessment. Respir Med. 2017 Apr;125:65-71. doi: 10.1016/j.rmed.2017.03.006. Epub 2017 Mar 6. PMID 28340864
- [Background] Rozanski C, Mura M. Multi-dimensional indices to stage idiopathic pulmonary fibrosis: a systematic review. Sarcoidosis Vasc Diffuse Lung Dis. 2014 Apr 18;31(1):8-18. PMID 24751449
- [Background] Hosein K, Le J, Mura M. Assessing the Therapeutic Response to Pirfenidone in Idiopathic Pulmonary Fibrosis: Can We Do Better than with Forced Vital Capacity Alone? Lung. 2017 Feb;195(1):101-105. doi: 10.1007/s00408-016-9963-3. Epub 2016 Nov 17. PMID 27858160
- [Background] Taha N, D'Amato D, Hosein K, Ranalli T, Sergiacomi G, Zompatori M, Mura M. Longitudinal functional changes with clinically significant radiographic progression in idiopathic pulmonary fibrosis: are we following the right parameters? Respir Res. 2020 May 19;21(1):119. doi: 10.1186/s12931-020-01371-7. PMID 32429952
- [Background] Hosein KS, Sergiacomi G, Zompatori M, Mura M. The CALIPER-Revised Version of the Composite Physiologic Index is a Better Predictor of Survival in IPF than the Original Version. Lung. 2020 Feb;198(1):169-172. doi: 10.1007/s00408-019-00295-4. Epub 2019 Dec 2. PMID 31792602
- [Background] Ley B, Ryerson CJ, Vittinghoff E, Ryu JH, Tomassetti S, Lee JS, Poletti V, Buccioli M, Elicker BM, Jones KD, King TE Jr, Collard HR. A multidimensional index and staging system for idiopathic pulmonary fibrosis. Ann Intern Med. 2012 May 15;156(10):684-91. doi: 10.7326/0003-4819-156-10-201205150-00004. PMID 22586007
- [Background] Wells AU, Desai SR, Rubens MB, Goh NS, Cramer D, Nicholson AG, Colby TV, du Bois RM, Hansell DM. Idiopathic pulmonary fibrosis: a composite physiologic index derived from disease extent observed by computed tomography. Am J Respir Crit Care Med. 2003 Apr 1;167(7):962-9. doi: 10.1164/rccm.2111053. PMID 12663338
- [Background] Jacob J, Bartholmai BJ, Rajagopalan S, Kokosi M, Nair A, Karwoski R, Raghunath SM, Walsh SL, Wells AU, Hansell DM. Automated Quantitative Computed Tomography Versus Visual Computed Tomography Scoring in Idiopathic Pulmonary Fibrosis: Validation Against Pulmonary Function. J Thorac Imaging. 2016 Sep;31(5):304-11. doi: 10.1097/RTI.0000000000000220. PMID 27262146
- [Background] du Bois RM, Weycker D, Albera C, Bradford WZ, Costabel U, Kartashov A, Lancaster L, Noble PW, Raghu G, Sahn SA, Szwarcberg J, Thomeer M, Valeyre D, King TE Jr. Ascertainment of individual risk of mortality for patients with idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2011 Aug 15;184(4):459-66. doi: 10.1164/rccm.201011-1790OC. PMID 21616999
- [Background] Flaherty KR, King TE Jr, Raghu G, Lynch JP 3rd, Colby TV, Travis WD, Gross BH, Kazerooni EA, Toews GB, Long Q, Murray S, Lama VN, Gay SE, Martinez FJ. Idiopathic interstitial pneumonia: what is the effect of a multidisciplinary approach to diagnosis? Am J Respir Crit Care Med. 2004 Oct 15;170(8):904-10. doi: 10.1164/rccm.200402-147OC. Epub 2004 Jul 15. PMID 15256390
- [Background] Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1384-7. doi: 10.1164/ajrccm.158.5.9710086. PMID 9817683
- [Background] Murciano D, Pichot MH, Boczkowski J, Sleiman C, Pariente R, Milic-Emili J. Expiratory flow limitation in COPD patients after single lung transplantation. Am J Respir Crit Care Med. 1997 Mar;155(3):1036-41. doi: 10.1164/ajrccm.155.3.9116983.
- [Background] Nathan SD, Shlobin OA, Barnett SD, Saggar R, Belperio JA, Ross DJ, Ahmad S, Saggar R, Libre E, Lynch JP 3rd, Zisman DA. Right ventricular systolic pressure by echocardiography as a predictor of pulmonary hypertension in idiopathic pulmonary fibrosis. Respir Med. 2008 Sep;102(9):1305-10. doi: 10.1016/j.rmed.2008.03.022. Epub 2008 Jul 10. PMID 18619825
- [Background] King TE Jr, Bradford WZ, Castro-Bernardini S, Fagan EA, Glaspole I, Glassberg MK, Gorina E, Hopkins PM, Kardatzke D, Lancaster L, Lederer DJ, Nathan SD, Pereira CA, Sahn SA, Sussman R, Swigris JJ, Noble PW; ASCEND Study Group. A phase 3 trial of pirfenidone in patients with idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2083-92. doi: 10.1056/NEJMoa1402582. Epub 2014 May 18. PMID 24836312
- [Background] Fischer A, Antoniou KM, Brown KK, Cadranel J, Corte TJ, du Bois RM, Lee JS, Leslie KO, Lynch DA, Matteson EL, Mosca M, Noth I, Richeldi L, Strek ME, Swigris JJ, Wells AU, West SG, Collard HR, Cottin V; "ERS/ATS Task Force on Undifferentiated Forms of CTD-ILD". An official European Respiratory Society/American Thoracic Society research statement: interstitial pneumonia with autoimmune features. Eur Respir J. 2015 Oct;46(4):976-87. doi: 10.1183/13993003.00150-2015. Epub 2015 Jul 9. PMID 26160873
- [Background] Khadawardi H, Mura M. A simple dyspnoea scale as part of the assessment to predict outcome across chronic interstitial lung disease. Respirology. 2017 Apr;22(3):501-507. doi: 10.1111/resp.12945. Epub 2016 Nov 8. PMID 27862639
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Wanger J, Clausen JL, Coates A, Pedersen OF, Brusasco V, Burgos F, Casaburi R, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson D, Macintyre N, McKay R, Miller MR, Navajas D, Pellegrino R, Viegi G. Standardisation of the measurement of lung volumes. Eur Respir J. 2005 Sep;26(3):511-22. doi: 10.1183/09031936.05.00035005. No abstract available. PMID 16135736
- [Background] Graham BL, Brusasco V, Burgos F, Cooper BG, Jensen R, Kendrick A, MacIntyre NR, Thompson BR, Wanger J. 2017 ERS/ATS standards for single-breath carbon monoxide uptake in the lung. Eur Respir J. 2017 Jan 3;49(1):1600016. doi: 10.1183/13993003.00016-2016. Print 2017 Jan. PMID 28049168
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Brennan P, Silman A. Statistical methods for assessing observer variability in clinical measures. BMJ. 1992 Jun 6;304(6840):1491-4. doi: 10.1136/bmj.304.6840.1491. No abstract available. PMID 1611375
- [Background] Slinker BK, Glantz SA. Multiple regression for physiological data analysis: the problem of multicollinearity. Am J Physiol. 1985 Jul;249(1 Pt 2):R1-12. doi: 10.1152/ajpregu.1985.249.1.R1. PMID 4014489
- [Background] Scrucca L, Santucci A, Aversa F. Regression modeling of competing risk using R: an in depth guide for clinicians. Bone Marrow Transplant. 2010 Sep;45(9):1388-95. doi: 10.1038/bmt.2009.359. Epub 2010 Jan 11. PMID 20062101
- [Background] Wang X, Ji X. Sample Size Estimation in Clinical Research: From Randomized Controlled Trials to Observational Studies. Chest. 2020 Jul;158(1S):S12-S20. doi: 10.1016/j.chest.2020.03.010. PMID 32658647
- [Background] Richeldi L, du Bois RM, Raghu G, Azuma A, Brown KK, Costabel U, Cottin V, Flaherty KR, Hansell DM, Inoue Y, Kim DS, Kolb M, Nicholson AG, Noble PW, Selman M, Taniguchi H, Brun M, Le Maulf F, Girard M, Stowasser S, Schlenker-Herceg R, Disse B, Collard HR; INPULSIS Trial Investigators. Efficacy and safety of nintedanib in idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2071-82. doi: 10.1056/NEJMoa1402584. Epub 2014 May 18. PMID 24836310
- [Background] Chambers DC, Yusen RD, Cherikh WS, Goldfarb SB, Kucheryavaya AY, Khusch K, Levvey BJ, Lund LH, Meiser B, Rossano JW, Stehlik J; International Society for Heart and Lung Transplantation. The Registry of the International Society for Heart and Lung Transplantation: Thirty-fourth Adult Lung And Heart-Lung Transplantation Report-2017; Focus Theme: Allograft ischemic time. J Heart Lung Transplant. 2017 Oct;36(10):1047-1059. doi: 10.1016/j.healun.2017.07.016. Epub 2017 Jul 19. No abstract available. PMID 28784324
- [Background] Kistler KD, Nalysnyk L, Rotella P, Esser D. Lung transplantation in idiopathic pulmonary fibrosis: a systematic review of the literature. BMC Pulm Med. 2014 Aug 16;14:139. doi: 10.1186/1471-2466-14-139. PMID 25127540
- [Background] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Background] Rajala K, Lehto JT, Sutinen E, Kautiainen H, Myllarniemi M, Saarto T. mMRC dyspnoea scale indicates impaired quality of life and increased pain in patients with idiopathic pulmonary fibrosis. ERJ Open Res. 2017 Dec 14;3(4):00084-2017. doi: 10.1183/23120541.00084-2017. eCollection 2017 Oct. PMID 29255720
- [Background] Nishiyama O, Taniguchi H, Kondoh Y, Kimura T, Kato K, Kataoka K, Ogawa T, Watanabe F, Arizono S. A simple assessment of dyspnoea as a prognostic indicator in idiopathic pulmonary fibrosis. Eur Respir J. 2010 Nov;36(5):1067-72. doi: 10.1183/09031936.00152609. Epub 2010 Apr 22. PMID 20413545
- [Background] Guyatt GH, Thompson PJ, Berman LB, Sullivan MJ, Townsend M, Jones NL, Pugsley SO. How should we measure function in patients with chronic heart and lung disease? J Chronic Dis. 1985;38(6):517-24. doi: 10.1016/0021-9681(85)90035-9. PMID 4008592
- [Background] Guyatt GH, Townsend M, Keller J, Singer J, Nogradi S. Measuring functional status in chronic lung disease: conclusions from a randomized control trial. Respir Med. 1989 Jul;83(4):293-7. doi: 10.1016/s0954-6111(89)80199-4. PMID 2692093
- [Background] Ora J, Calzetta L, Pezzuto G, Senis L, Paone G, Mari A, Portalone S, Rogliani P, Puxeddu E, Saltini C. A 6MWT index to predict O2 flow correcting exercise induced SpO2 desaturation in ILD. Respir Med. 2013 Dec;107(12):2014-21. doi: 10.1016/j.rmed.2013.10.002. Epub 2013 Oct 10. PMID 24161677
- [Background] du Bois RM, Weycker D, Albera C, Bradford WZ, Costabel U, Kartashov A, Lancaster L, Noble PW, Sahn SA, Szwarcberg J, Thomeer M, Valeyre D, King TE Jr. Six-minute-walk test in idiopathic pulmonary fibrosis: test validation and minimal clinically important difference. Am J Respir Crit Care Med. 2011 May 1;183(9):1231-7. doi: 10.1164/rccm.201007-1179OC. Epub 2010 Dec 3. PMID 21131468
- [Background] Lama VN, Flaherty KR, Toews GB, Colby TV, Travis WD, Long Q, Murray S, Kazerooni EA, Gross BH, Lynch JP 3rd, Martinez FJ. Prognostic value of desaturation during a 6-minute walk test in idiopathic interstitial pneumonia. Am J Respir Crit Care Med. 2003 Nov 1;168(9):1084-90. doi: 10.1164/rccm.200302-219OC. Epub 2003 Aug 13. PMID 12917227
- [Background] Zappala CJ, Latsi PI, Nicholson AG, Colby TV, Cramer D, Renzoni EA, Hansell DM, du Bois RM, Wells AU. Marginal decline in forced vital capacity is associated with a poor outcome in idiopathic pulmonary fibrosis. Eur Respir J. 2010 Apr;35(4):830-6. doi: 10.1183/09031936.00155108. Epub 2009 Oct 19. PMID 19840957
- [Background] King TE Jr, Safrin S, Starko KM, Brown KK, Noble PW, Raghu G, Schwartz DA. Analyses of efficacy end points in a controlled trial of interferon-gamma1b for idiopathic pulmonary fibrosis. Chest. 2005 Jan;127(1):171-7. doi: 10.1378/chest.127.1.171. PMID 15653980
- [Background] Lee SH, Park JS, Kim SY, Kim DS, Kim YW, Chung MP, Uh ST, Park CS, Park SW, Jeong SH, Park YB, Lee HL, Shin JW, Lee EJ, Lee JH, Jegal Y, Lee HK, Kim YH, Song JW, Park MS. Comparison of CPI and GAP models in patients with idiopathic pulmonary fibrosis: a nationwide cohort study. Sci Rep. 2018 Mar 19;8(1):4784. doi: 10.1038/s41598-018-23073-3. PMID 29555917
- [Background] Salisbury ML, Xia M, Zhou Y, Murray S, Tayob N, Brown KK, Wells AU, Schmidt SL, Martinez FJ, Flaherty KR. Idiopathic Pulmonary Fibrosis: Gender-Age-Physiology Index Stage for Predicting Future Lung Function Decline. Chest. 2016 Feb;149(2):491-498. doi: 10.1378/chest.15-0530. Epub 2016 Jan 12. PMID 26425858
- [Background] Levine GN, McCullough KP, Rodgers AM, Dickinson DM, Ashby VB, Schaubel DE. Analytical methods and database design: implications for transplant researchers, 2005. Am J Transplant. 2006;6(5 Pt 2):1228-42. doi: 10.1111/j.1600-6143.2006.01277.x. PMID 16613598
- [Background] Lyu DM, Goff RR, Chan KM. The Lung Allocation Score and Its Relevance. Semin Respir Crit Care Med. 2021 Jun;42(3):346-356. doi: 10.1055/s-0041-1729541. Epub 2021 May 24. PMID 34030198
- [Derived] Manzetti GM, Hosein K, Cecchini MJ, Kwan K, Abdelrazek M, Zompatori M, Rogliani P, Mura M. Validation of the risk stratification score in idiopathic pulmonary fibrosis: study protocol of a prospective, multi-centre, observational, 3-year clinical trial. BMC Pulm Med. 2021 Dec 4;21(1):396. doi: 10.1186/s12890-021-01753-7. PMID 34863146